CLINICAL TRIAL: NCT04164849
Title: Extracorporeal Photopheresis of Patients With Crohn's Disease Using 5-aminolevulinic Acid
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Jørgen Jahnsen, Professor, University Hospital, Akershus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: twostepala
Record Dates: First submitted 2019-11-08; First posted 2019-11-15 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Crohn Disease
Keywords: Crohns Disease; Photopheresis; 5-aminolevulinic acid; Gliolan; UVA-PIT
MeSH Terms: conditions — Crohn Disease | interventions — Aminolevulinic Acid; Blood Transfusion

STUDY DESIGN:
Intervention Model Description: A combined phase 1/2 pilot study with emphasize on safety/tolerability but also clinical efficacy/effect
Masking Description: all patients will receive active treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 5-ALA photopheresis (Experimental): All patients will receive 5-aminolevulinic acid (5-ALA) in combination with blue light photopheresis. The investigators will collect mononuclear cells by connecting patient to Spectra Optia with CMNC (continuous mononuclear cell collection protocol), and these cells will include active T-lymphocytes. 5-ALA will be incubated for 1 hour to produce photoactive protoporphyrin-IX (PpIX) before light exposure.
  Interventions: Drug: 5-aminolevulinic acid; Procedure: Blue light photopheresis; Procedure: Transfusion; Procedure: Continuous Mononuclear Cell Collection (CMNC)

INTERVENTIONS:
Drug: 5-aminolevulinic acid — 5-aminolevulinic acid (30 mg/ml) will be added to mononuclear cells in a dose of 3 millimolar and incubated for 1 hour
Procedure: Blue light photopheresis — The mononuclear cells incubated with 5-aminolevulinic acid for 1 hour will be exposed to blue light.
Procedure: Transfusion — The treated cells are transferred back to the patient as a standard blood transfusion
Procedure: Continuous Mononuclear Cell Collection (CMNC) — The mononuclear cells are collected using the Spectra Optia with the Continuous Mononuclear Cell Collection protocol. 90 ml of mononuclear cells will be collected and 100 ml of 0,9% saline will be added to dilute the cells before incubation with drug and photopheresis.

SUMMARY:
In the clinical trial the investigators will assess efficacy, safety and tolerability after single and multiple doses of 3 millimolar 5 aminolevulinic acid (Gliolan®) in combination with blue-light (405 nanometer) photopheresis in patients with active crohns disease. The study is a proof-of-concept pilot with up to 10 included patients where every patient will get active treatment. The use of 5-aminolevulinic acid in combination with blue-light photopheresis is a first-in-human trial. Primary endpoints include clinical response and adverse events (safety). Secondary endpoints include endoscopic improvement, quality of life questionnaires, faecal calprotectin, C-reactive protein and mechanisms of action (differences in t-cells and other cells before and after treatment). All patients will get treatment every 2 weeks for 10 weeks (6 treatments-induction) with evaluation at week 13. If any effect on week 13 eligible for study extension with treatment every 4 weeks for up to 12 months for the first 5 patients. The latter 5 patients will be referred to standard of care on the week 13 visit. Through the study the investigators will see if this kind of photopheresis is safe and can be an option for a larger randomized-controlled-trial. In addition the investigators will see if photopheresis as an option can be further developed for other diseases as well (ie other T-cell mediated diseases or patients already receiving photopheresis as a treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Age above 18
3. Male or female patient with active Crohn's disease (6)
4. Women of childbearing potential (WOCBP) will have to use highly effective methods of contraception throughout the entire study.
5. Inadequate response (a) or intolerance to biological therapy

   a. Inadequate response on ongoing treatment is defined as: i. Progressive disease: increasing Harvey Bradshaw Index/Calprotectin/Simple Endoscopic Score for Crohns Disease and/or worsening of radiologic images after 6 months.

   ii. Stable disease: no-response after 6 months
6. Active inflammation in the gut documented by

   1. Harvey Bradshaw Index >5 and
   2. Endoscopy with Simple Endoscopic Score for Crohns Disease equal to or above 6 points or equal to or above 4 points if only isolated ileitis is present and/or
   3. Inflammatory marker; fecal calprotectin > 250 and/or C reactive protein > 5

Exclusion Criteria:

1. Photosensitive comorbidities, porphyria or known hypersensitivity to 5-aminolevulinic acid or porphyrins
2. Patients with aphakia
3. Pregnant or breast-feeding women. A negative urine pregnancy test must be demonstrated in female patients of child-bearing potential at the Screening Visit and before every treatment.
4. Ongoing cardiac and pulmonary diseases or aspartate transaminase alanine aminotransferase, Bilirubin or International Normalized Ratio value ≥ 3x upper limit of normal or clinically significant electrocardiogram findings
5. Subjects with polyneuropathy
6. Uncontrolled infection or fever
7. History of heparin-induced thrombocytopenia, absolute neutrophil count <1x109, platelet count <20x10 9
8. Body weight below 40 kg
9. Investigator considers subject unlikely to comply with study procedures, restrictions and requirements.
10. Presence of other gastrointestinal diseases potentially influencing the study endpoints
11. History of any clinically significant disease or disorder which in the opinion of the investigator, may either put the patient at risk because of participation in the study, or influence the result or the patient's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Clinical response | Week 13, 26 (28 for patients not eligible for study extension and the latter 5 patients), 38, 50, 64 and 3 months after last treatment
  Clinical response (Harvey Bradshaw Index change > 3 from baseline or less than 4 points)
Safety and tolerability adverse events | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Frequency, seriousness and intensity of adverse events
Safety and tolerability Electrocardiogram-PR interval | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in PR interval before and after treatment
Safety and tolerability Electrocardiogram-PR segment | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in PR segment before and after treatment
Safety and tolerability Electrocardiogram-QT interval | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in QT interval before and after treatment
Safety and tolerability Electrocardiogram-ST segment | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in ST segment before and after treatment
Safety and tolerability Electrocardiogram-T wave | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in T wave before and after treatment
Safety and tolerability Electrocardiogram-QRS complex | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in QRS complex before and after treatment
Safety and tolerability vital signs | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Vital signs (heart rate) before and after treatment
Safety and tolerability blood pressure | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Vital signs (systolic and diastolic blood pressure) before and after treatment
Alkaline phosphatase | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in serum alkaline phosphatase (U/L) before and after treatment
Aspartate transferase | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in serum aspartate transferase(U/L) before and after treatment
Alanine aminotransferase | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in serum alanine aminotransferase (U/L) before and after treatment
Albumin | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Serum Albumin (g/L) before and after treatment
Bilirubin | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Serum Bilirubin (micromol/L) before and after treatment
Gamma glutamyltransferase | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Serum gamma glutamyltransferase (U/L) before and after treatment
White cell count | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Blood White cell count (10^9/L) before and after treatment
Neutrophil granulocytes | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Blood neutrophil granulocytes (10^9/L) before and after treatment
Lymphocytes | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Blood Lymphocytes (10^9/L) before and after treatment
Monocytes | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Blood Monocytes (10^9/L) before and after treatment
Eosinophile granulocytes | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Blood Eosinophile granulocytes (10^9/L) before and after treatment
Basophile granulocytes | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Blood Basophile granulocytes (10^9/L) before and after treatment
Platelet count | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Blood Platelet count (10^9/L) before and after treatment
Mean Cell Volume | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Blood Mean Cell Volume (fL) before and after treatment
Mean Cell hemoglobin | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Blood Mean Cell hemoglobin (picogram) before and after treatment
International Normalized Ratio | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Blood International Normalized Ratio (0,8-1,2) before and after treatment
Hemoglobin | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Blood Hemoglobin (g/dL) before and after treatment
Calcium | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Serum Calcium (millimol/L) before and after treatment
Potassium | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Serum Potassium (millimol/L) before and after treatment
Sodium | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Serum Sodium (millimol/L) before and after treatment
Creatinin | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Serum Creatinine (micromol/L) before and after treatment
Lactate Dehydrogenase | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Serum Lactate Dehydrogenase (U/L) before and after treatment
Cholesterol | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Serum Cholesterol (millimol/L) before and after treatment
Total Protein | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Serum Total Protein (g/L) before and after treatment
Carbamide | Before every treatment visit (every second week from week 0-10, every 4th week from week 14-62, week 28 for patients not eligible for study extension and latter 5 patients) in addition to week 64 and 3 months after last treatment.
  Changes in Serum Carbamide (millimol/L) before and after treatment

SECONDARY OUTCOMES:
CD4+ and CD8+ T cell subpopulations | Week 0, 10 (all patients) and 50 (patients of the first 5 subjects eligible for study extension)
  Number of CD4+ and CD8+ T cell subpopulations before and after treatment assessed by flow cytometry.
Apoptosis and necrosis | Week 0, 10 (all patients) and 50 (patients of the first 5 subjects eligible for study extension)
  Number of cells in apoptosis or necrosis before and after treatment assessed by flow cytometry
Clinical remission | Week 13 and/or sustained/delayed response in week 26 (28 for patients not eligible for study extension and the latter 5 patients), 38, 50, 64 and 3 months after last treatment.
  Harvey Bradshaw Index < 5 points
Endoscopic efficacy | Week 13 (all patients) and 64 (patients of the first 5 subjects eligible for study extension) with baseline visit as reference.
  Simple Endoscopic Score for Crohns Disease >49 % improvement or < 3 (endoscopic remission)
Faecal calprotectin | Week 13, 26 (28 for patients not eligible for study extension and the latter 5 patients), 38, 50, 64 and/or 3 months after last treatment
  Change from baseline
Concentration of C reactive protein in blood | Week 13, 26 (28 for patients not eligible for study extension and the latter 5 patients), 38, 50, 64 and/or 3 months after last treatment
  Change from baseline
Quality of life questionnaire Short-Form 36 (SF-36) | Week 13, 26 (28 for patients not eligible for study extension and the latter 5 patients), 38, 50, 64 and/or 3 months after last treatment
  Change of both total and subscores of SF-36 from baseline. Min 0 Max 100. Higher value is better quality of life.
Quality of life questionnaire Inflammatory Bowel Disease Questionnaire (IBDQ) | Week 13, 26 (28 for patients not eligible for study extension and the latter 5 patients), 38, 50, 64 and/or 3 months after last treatment
  Change of both total and subscores of IBDQ from baseline. Min 32 Max 224. Higher value is better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Akershus University Hospital, Lorenskog, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No